CLINICAL TRIAL: NCT06561217
Title: Assessing the Performance of Artificial Intelligence (AI)-Augmented Electronic Health Record (EHR) Data Abstraction for Clinical Trial Patient Screening
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: Mendel AI (Industry)
Responsible Party: Sponsor
Other Study IDs: 854016
Record Dates: First submitted 2024-08-16; First posted 2024-08-19 (Actual); Results first posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- AI-alone
  Interventions: Other: Chart review
- Human-alone
  Interventions: Other: Chart review
- Human + AI
  Interventions: Other: Chart review

INTERVENTIONS:
Other: Chart review — Chart review

SUMMARY:
Identifying eligible patients is a key process in the clinical trial enterprise. Currently, this process relies on time-intensive manual chart review, creating a rate-limiting step for trial participation. The integration of AI technology into the trial screening process has potential to improve participation rates. This study aims to assess the performance (accuracy, efficiency) of AI-augmented patient identification and inform optimal integration into clinical research screening processes.

DETAILED DESCRIPTION:
The objective of this study is to assess and compare the accuracy and efficiency of three different approaches to abstracting clinical data used to identify oncology patients who meet the inclusion criteria for participation in clinical trials. The three approaches under evaluation include: (1) an autonomous AI algorithm (Mendel AI; developed by artificial intelligence startup company Mendel) which analyzes patient medical records to extract relevant clinical facts ("AI-alone"); (2) a human researcher who manually reviews patient charts as per the current norm/practice ("Human-alone"); and (3) a human researcher utilizing AI augmentation ("Human+AI"), where Mendel AI serves as a supportive tool in the decision-making process by providing the researcher a list of elements abstracted by the AI algorithm and a rank-order list of patients most likely to meet inclusion criteria for a trial.

The study primarily aims to compare (1) the chart-level accuracy of the Human+AI collaboration relative to Human-alone given the relevance of this comparison for real-world clinical workflows, defined by the percentage of pre-identified chart elements classified correctly compared against a predetermined "gold standard"; and (2) the efficiency of the Human+AI vs. Human-alone arms, defined by the time per chart review in minutes, measured for each chart.

Our hypotheses are (1) the Human+AI arm will be non-inferior in accuracy when compared to the Human-alone arm, in relation to a predetermined "gold standard", and (2) that a Human+AI arm will be superior in efficiency of abstraction when compared to Human-alone screening.

The identification of eligible patients for clinical trials is a critical component of clinical research, as it directly impacts patient recruitment, study enrollment, and the generalizability of research findings. Currently, the process of identifying eligible patients often relies on manual chart review by clinical research staff, which can be time-consuming, labor-intensive, and prone to human error. Consequently, eligible patients may be overlooked, and opportunities for trial participation may be missed. The integration of AI technology into the patient identification process has the potential to enhance the accuracy and efficiency of this critical task, leading to improved clinical trial recruitment and outcomes.

This study holds important implications for the field of clinical research by evaluating the effectiveness of AI-augmented patient identification compared to traditional manual methods and autonomous AI algorithms. By examining the strengths and limitations of each approach, the study will provide valuable insights into the optimal integration of AI technology in clinical research processes. Furthermore, the results of this study have the potential to benefit patients by improving their access to clinical trials and increasing awareness of available treatment options. For clinical research institutions, enhancing the efficiency of patient identification can lead to more effective use of research resources and the potential for accelerated clinical trial timelines. Ultimately, the findings of this study may contribute to advancements in clinical research practices, promoting more equitable access to trials and facilitating the development of innovative treatments for patients with cancer.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of colorectal or non-small cell lung cancer.
* A minimum of 5 patient documents in the Mendel database.
* Most recent document was within 5 years from the time of data extraction.

Exclusion Criteria:

* None.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: De-identified patient charts from community oncology practices, with a diagnosis of non-small cell lung cancer (NSCLC) or colorectal cancer (CRC).
Sampling Method: Probability Sample
Enrollment: 355 (Actual)
Dates: Start 2023-08-18 (Actual); Primary Completion 2024-07-12 (Actual); Study Completion 2024-07-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Emory University, Atlanta, Georgia
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared.

REFERENCES:
- [Derived] Parikh RB, Kolla L, Beothy EA, Ferrell WJ, Laventure B, Guido M, Girard A, Li Y, Dosoky KEM, Tarabishy K, Patel PS, Andalcio A, Maloney K, Mena JU, Salloum W, Chen J, Emanuel EJ. Human-AI teaming to improve accuracy and efficiency of eligibility criteria prescreening for oncology trials: a randomized evaluation trial using retrospective electronic health records. Nat Commun. 2026 Feb 3. doi: 10.1038/s41467-026-68873-8. Online ahead of print. PMID 41634037

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Each record will be reviewed via all 3 arms, so the total enrollment will be 355.
Groups:
- All Participants: Patients that underwent all chart reviews (Human-alone, AI-alone, and Human + AI)
Period: Human-alone
Arm/Group | All Participants
Started | 355
Completed | 355
Not Completed | 0
Period: AI-alone
Arm/Group | All Participants
Started | 355
Completed | 355
Not Completed | 0
Period: Human + AI
Arm/Group | All Participants
Started | 355
Completed | 355
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Each participated in all 3 arms, for an overall total of 355.
Groups:
- All Participants: Patients who underwent Human-alone, AI-alone, and Human+AI chart review
Arm/Group | All Participants
Number analyzed (Participants) | 355
Age, Customized [Count of Participants; unit: Participants]
  <18 years | 0
  ≥18 years | 355
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Sex/gender were not collected from any participant.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 355
Cancer Type [Count of Participants; unit: Participants]
  Non-Small Cell Lung Cancer | 195
  Colorectal Cancer | 160

OUTCOME MEASURES:

1. Primary Outcome: Abstracted Chart-level Accuracy
Description: The primary outcome measured was mean chart-level accuracy, defined as the percentage of elements identified by clinical research coordinators among all elements in the gold-standard set, measured for each chart, and averaged across all charts. Research coordinator-abstracted responses were identified as being accurate when they exactly matched with the gold-standard set. The gold-standard set was determined by 2-3 clinicians blinded to experimental arms.
Time Frame: 1 year
Population: The study population was drawn from a 15-physician community oncology practice in California serving patients from urban and surrounding rural communities. This study cohort consisted of unstructured medical records from patients within the dataset with 1) a diagnosis of non-small cell lung cancer (NSCLC) or colorectal cancer (CrCa), 2) a minimum of five clinical documents available, and 3) the most recent document being within five years from the time of data extraction.
Measure: Mean (Standard Deviation); unit: % of elements correctly abstracted
Groups:
- Human + AI: Charts reviewed by AI-augmented human reviewers
- Human-alone: Charts reviewed by human abstraction alone - no AI support.
- AI-alone: Charts reviewed by AI model alone, without Human support
Arm/Group | Human + AI | Human-alone | AI-alone
Number analyzed (Participants) | 355 | 355 | 355
% of elements correctly abstracted | 76.10 (20.59) | 71.48 (24.92) | 59.92 (23.75)
Statistical Analysis 1: Comparison: Human + AI vs Human-alone; A Shapiro-Wilk test was used to assess normality of paired differences in chart-level accuracy (alpha = 0.05). A one-sided, paired Wilcoxon Rank Sum test (alpha = 0.05) was employed to test the primary null hypothesis of whether chart-level accuracy of the Human+AI arm for EHR chart abstraction was non-inferior to the chart-level accuracy of a Human-alone arm abstraction by at least 5% (i.e., noninferiority margin); Test type: Non-Inferiority — A predefined non-inferiority margin of 0.05 was used. The primary study was powered on a retrospective, paired, non-inferiority design to evaluate abstraction accuracy of elements commonly used to help screen patients for clinical trials; p < 0.001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.02, 95% CI 1-sided [lower limit 0.00007515] — The upper bound of the 95% confidence interval is Inf due to the test being one-sided. Alternative hypothesis: true median location shift is greater than -0.05
Statistical Analysis 2: Comparison: Human + AI vs Human-alone; A Shapiro-Wilk test was used to assess normality of paired differences in chart-level accuracy (alpha = 0.05). A one-sided, paired Wilcoxon Rank Sum test (alpha = 0.05) was employed to test the null hypothesis of whether chart-level accuracy of the Human+AI arm for EHR chart abstraction was superior to the chart-level accuracy of a Human-alone arm abstraction; Test type: Superiority — The primary study was powered on a retrospective, paired, superiority design to evaluate abstraction accuracy of elements commonly used to help screen patients for clinical trials; p = 0.002, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.02

2. Secondary Outcome: Efficiency of Chart-level Abstraction (in Minutes)
Description: Efficiency was calculated as the number of minutes spent on each chart abstraction.
Time Frame: 1 year
Population: The study population was the same as the study population described in the primary outcome analysis population description section. However, AI-alone chart reviews were NOT analyzed for efficiency. Data for the secondary outcome of efficiency was not collected for the AI-alone arm and therefore cannot be reported in the outcome table. This was prespecified, as its fully automated nature renders direct comparison with human-involved workflows inappropriate and uninformative.
Measure: Median (Inter-Quartile Range); unit: Number of minutes spent on abstraction
Arm/Group | Human + AI | Human-alone
Number analyzed (Participants) | 355 | 355
Number of minutes spent on abstraction | 32.12 [20.55 to 48.67] | 31.75 [20.27 to 49.34]
Statistical Analysis 1: Comparison: Human + AI vs Human-alone; A two-sided, paired Wilcoxon Rank Sum test (alpha = 0.05) was employed to test for difference between chart-level efficiency of the Human+AI arm and chart-level efficiency of the Human-alone arm abstraction; Test type: Equivalence — Null hypothesis: True difference is equal to 0. Alternate hypothesis: true difference is not equal to 0; p = 0.513, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.66, 95% CI 2-sided [-1.25 to 2.55]

ADVERSE EVENTS:
Time Frame: Not applicable. Adverse events were not collected.
Description: Not applicable. Adverse events were not collected.
Arm/Group | AI-alone | Human-alone | Human + AI
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-01-23): https://cdn.clinicaltrials.gov/large-docs/17/NCT06561217/Prot_SAP_000.pdf